CLINICAL TRIAL: NCT07041164
Title: Diagnostic Performance and Children's Acceptance of Near-Infrared Light Transillumination and Bitewing Radiographs for Detecting Proximal Cavitation in Primary Molars of Patients Aged 4 to 10 Years
Acronym: NILT
Status: Recruiting | Type: Observational
Sponsor: Sawanya Prutthithaworn (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor-Investigator, Sawanya Prutthithaworn, Dr, Mahidol University
Organization: Mahidol University (Other)
Other Study IDs: MU-DT/PY-IRB 2025/025.0304
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dental Caries (Diagnosis); Diagnostic Imaging; Optical Imaging; Radiographic Image Interpretation, Computer-Assisted; Proximal Dental Caries; Tooth, Deciduous
Keywords: proximal caries; primary molars; Pediatric Patients; Bitewing Radiography; Near-Infrared Light Transillumination; DIAGNOcam; clinical cavitation; children acceptance; Diagnostic accuracy
MeSH Terms: conditions — Dental Caries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- 4-6 years old
  Interventions: Diagnostic Test: Bitewing radiograph; Diagnostic Test: Near-infrared light transillumination
- 6-8 years old
  Interventions: Diagnostic Test: Bitewing radiograph; Diagnostic Test: Near-infrared light transillumination
- 8-10 years old
  Interventions: Diagnostic Test: Bitewing radiograph; Diagnostic Test: Near-infrared light transillumination

INTERVENTIONS:
Diagnostic Test: Bitewing radiograph — Digital radiograph, proximal caries, initial caries
Diagnostic Test: Near-infrared light transillumination — DIAGNOcam, proximal caries, initial caries

SUMMARY:
The goal of this observational study is to compare the diagnostic performance of three detection methods for approximal carious lesions in primary molars among pediatric patients aged 4-10 years. The study focuses on children in three age groups: 4-6 years, 6-8 years, and 8-10 years. The main questions it aims to answer are:

* Are the sensitivity, specificity, accuracy, and area under the curve (AUC) different across the three diagnostic techniques (bitewing radiography, near-infrared light transillumination, and their combination)?
* Are these diagnostic parameters influenced by patient age?
* Which technique yields the highest level of patient acceptance?

Researchers will compare the three diagnostic approaches to determine whether age influences diagnostic performance and patient acceptance.

Participants will:

* Be examined using bitewing radiography and near-infrared light transillumination
* Undergo tooth separation for 7 days using orthodontic elastic separators
* Receive clinical examination of the target approximal surface
* Be asked to rate their experience using the Simplified Facial Pain Scale (S-FPS)

DETAILED DESCRIPTION:
* 58 carious lesions classified as RA2 and RA3 according to the ICDAS II criteria from three groups of 4-6 years, 6-8 years, and 8-10 years pediatric patients will be examined by near-infrared light transillumination
* The patient acceptance towards bitewing radiograph and near-infrared light transillumination will be evulated by Simplified Facial Pain Scale (S-FPS)
* Diagnostic performance will be assessed by calculating sensitivity, specificity, accuracy, and the area under the curve (AUC)
* The diagnostic efficacy of the caries detection methods will be analyzed using repeated measures ANOVA, and patient acceptance will be assessed using the Chi-square test, with statistical significance set at p < 0.05 and a 95% confidence level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children aged 4-10 years
* Low risk for periodontal disease
* At least one quadrant contains fully erupted, well-aligned adjacent primary molars that are free of restorations, exhibit no clinically visible cavitated caries, demonstrate tooth mobility of grade 2 or less, show no developmental dental anomalies
* Bitewing radiographs show at least one radiolucent lesion in the proximal surface of a primary molar classified as RA2 or RA3 according to the ICDAS II radiographic criteria

Exclusion Criteria:

* Root resorption exceeding two-thirds of the root length
* Demonstrate Frankl's behavior rating scale of 1 during either near-infrared light transillumination examination or tooth separation

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric dental clinic
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis performance | From enrollment to clinical examination on day 7th
  The diagnostic performance will be described by sensitivity, specificity, accuracy, and the Area Under the Curve (AUC), with values ranging from 0 to 1 for each parameter.
  * For sensitivity, zero is equivalent to no true positives detected, and 1 indicates all true positives detected
  * For specificity, zero is equivalent to no true negatives detected, and 1 indicates all true negatives detected
  * For accuracy, zero is equivalent to all cases misclassified, and 1 indicates all cases correctly classified
  * For AUC, zero is equivalent to a perfectly incorrect classification, and 1 indicates a perfectly correct classification
Age-influenced on diagnostic performance | From enrollment to clinical examination at day 7th
  The diagnostic performance for each age group will be described by sensitivity, specificity, accuracy, and the Area Under the Curve (AUC), with values ranging from 0 to 1 for each parameter.
  * For sensitivity, zero is equivalent to no true positives detected, and 1 indicates all true positives detected.
  * For specificity, zero is equivalent to no true negatives detected, and 1 indicates all true negatives detected.
  * For accuracy, zero is equivalent to all cases misclassified, and 1 indicates all cases correctly classified.
  * For AUC, zero is equivalent to a perfectly incorrect classification, and 1 indicates a perfectly correct classification.

SECONDARY OUTCOMES:
Children's acceptance | From enrollment to examination at day 0
  Children's acceptance will be evaluated using the Simplified Facial Pain Scale (S-FPS), which ranges from 0 to 10. The minimum value is 0, representing "no pain", and the maximum value is 10, representing "severe pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Hospital, Faculty of Dentistry, Mahidol University (Phayathai Campus), Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD), as required by the ethical approval granted by MU-DT/PY-IRB, will remain confidential and will not be disclosed. All data will be reported in aggregate form in publications or reports, ensuring that no individual participant can be identified. Any disclosure beyond these conditions will require an amendment to the approved ethical protocol.